# HİJYENİK PED AMBALAJI ÜZERINDEKİ YAZILI VE GÖRSEL MESAJLARIN KADINLARIN AİLE PLANLAMASINA İLIŞKİN BİLGİ VE TUTUMLARINA ETKİSİ: RANDOMİZE KONTROLLÜ ÇALIŞMA YÖNTEM

Bu çalışmanın, randomize kontrollü deneysel bir çalışma olarak 01 Ocak 2024- 01 Ocak 2025 tarihleri arasında yapılması planlanmıştır. Randomize kontrollü çalışma; yeni çıkan bir ilacı, bir tedaviyi veya başka bir müdahale çeşidini test etmek amacıyla benzer özelliklere sahip kişilerin deney ve kontrol grubuna ayrıldığı çalışma modelidir. Araştırmanın evrenini, Samsun İl Sağlık Müdürlüğü'nün Atakum ilçesinde bulunan Aile Sağlık Merkez'lerine (ASM) (18 ASM) bebeğinin bakım ve takibi için gelen kadınlar oluşturacaktır. Araştırmanın örneklemi, müdahale grubu ve kontrol grubu olmak üzere iki gruba ayrılacaktır. Araştırmada örneklem hacminin hesaplanması, Özer ve Yaman-Sözbir (2022)'in kontrasepsiyon eğitiminde kullanılan mizahın üniversite öğrencilerinin kontraseptif yöntemlere ilişkin tutumlarına etkisini değerlendirdiği çalışmaya dayalı olarak yapılmıştır. Deney grubunun Aile Planlamasına Yönelik Tutum Ölçeği son test ortalama ve standart sapma değeri 148,14±15,29, kontrol grubunun Aile Planlamasına Yönelik Tutum Ölçeği son test ortalama ve standart sapma değeri 138,29±14,64'dür. İlgili makalenin ortalama ve standart sapma değerleri G\*Power 3.1.9.2 programında bağımsız gruplarda t-testi kullanılarak effect size: 0,65 olarak hesaplanmıstır. Bu arastırmanın örneklemine alınması gereken en az birey sayısı G\*Power 3.1.9.2 ile effect size: 0.65,  $\alpha = 0.05$ , power: 0.80 alınarak hesaplanmış ve örneklem hacmi 78 (müdahale grubu: 39, kontrol grubu: 39) olarak belirlenmiştir. Araştırmanın analiz gücünü arttırmak için örneklem hacmini %30 artırarak olasılıksız örnekleme (gelişi güzel) yöntemi ile toplamda 100 kişinin alınması planlanmıştır (müdahale grubu: 50 ve kontrol grubu: 50). Müdahale grubu ve kontrol grubunda yer alan kadınlar eğitim düzeyi bakımından tabaka oluşturulacak ve grupların homojen dağılımı sağlanacaktır. Katılımcıların hangi grupta yer alacağı rastgele sayı üretme programı "Random Team Generator" adlı web sitesi üzerinden tam randomizasyon tekniğiyle belirlenecektir.

**t tests** - Means: Difference between two independent means (two groups)

= 1

Analysis: A priori: Compute required sample size

Input: Tail(s) = Two

Effect size d = 0.65  $\alpha$  err prob = 0.05

Power (1- $\beta$  err prob) = 0.80

Allocation ratio N2/N1

Output: Noncentrality parameter  $\delta$  = 2.8703223 Critical t = 1.9916726

Df = 76
Sample size group 1 = 39
Sample size group 2 = 39
Total sample size = 78
Actual power = 0.8089174



# Çalışmaya Alınma Kriterleri

- > 18-49 yaş aralığında,
- En az ilkokul mezunu olan,
- > 9-18 aylık bebeği olan,
- > AP yöntemi kullanmayan veya geleneksel AP yöntemleri (geri çekme, takvim yöntemi),
- > Evli ve cinsel partneri mevcut olan,
- Aktif cinsel yaşamı olan,
- > Düzenli menstrual siklusu olan,
- iletişimi engelleyen herhangi bir engeli olmayan,
- > Telefon numarasını vermeye gönüllü olan,
- > Akıllı telefon kullanan.
- En az ilkokul mezunu olan kadınlar dahil edilecektir.

#### Çalışmaya Alınmama Kriterleri

- Doğum sonu dönemde aile planlaması eğitimi alan,
- > Modern AP yöntemlerini kullanan,
- > Doğum sonu dönemde kanama gibi komplikasyonlardan dolayı histerektomi ameliyatı uygulanan,
- infertilite öyküsü olan ve yardımcı üreme teknikleri ile gebe kalmış olan,
- Menstrual siklusu olumsuz etkileyen herhangi bir sağlık sorunu (tiroid, kanser gibi) olan,
- ➤ Cinsel sağlığı olumsuz etkileyen herhangi bir kronik hastalık (kanser, diabet, hipertansiyon, hiperkolesterolemi, kalp hastalığı vb.) ya da ilaç (diüretik, antihipertansif, antihistaminik, antikolinerjik vb.) kullanımı olan,
- > Gebelik olan ya da tekrar gebelik planlayan,

Araştırmaya katılmayı kabul etmeyen ya da araştırmaya katılmaktan vazgeçme, yanlış ya da eksik bilgi veren kadınlar araştırmaya dahil edilmeyecektir.

# Veri Toplama Araçları

Araştırmada Kişisel Bilgi Formu ve Aile Planlaması Tutum Ölçeği kullanılacaktır.

Kişisel Bilgi Formu: Bu form, araştırmacılar tarafından literatür incelenerek oluşturulmuştur (Gavas ve İnal, 2017; Yağmur ve Keskin, 2019; Nazik ve ark, 2021; Özer ve Yaman-Sözbir, 2022). Form iki bölüm ve toplam 47 sorudan oluşmaktadır. Formun birinci bölümünde kadınların sosyodemografik özelliklerini sorgulayan 8 soru (yaş, aile tipi, eğitim düzeyi gibi), menstrual siklus özelliklerini sorgulayan 3 soru (en son menstrual kanama zamanı, menstrual kanama süresi ve menstrual siklusu), obstetrik özelliklerini sorgulayan 11 soru (gebelik sayısı gibi) ve aile planlaması kullanımı ile ilgili özelliklerini sorgulayan 10 soru (herhangi bir aile planlaması yöntemi kullanıma durumu, kullanılan aile planlaması yöntemi gibi) olmak üzere toplam 32 sorudan oluşmaktadır. Formun ikinci bölümünde (ikinci görüşmede doldurulacaktır) kadınların aile planlaması kullanımı ile ilgili özelliklerini sorgulayan 11 soru (herhangi bir aile planlaması yöntemi kullanıma durumu, kullanılan aile planlaması yöntemi gibi) ve hijyenik ped ambalajı ile ilgili düşünceleri sorgulayan 5 soru (hijyenik ped kullanılan dönemde ambalaj üzerindeki mesajları okuma durumu, hijyenik pedlerin yaygınlaştırılması halinde aile planlaması ile ilgili farkındalık yaratacağı düşüncesi gibi) olmak üzere toplam 16 sorudan oluşmaktadır. Formun birinci ve ikinci bölümünde toplam 48 soru yer almaktadır.

Aile Planlaması Bilgi Formu: Bu form, araştırmacılar tarafından literatür incelenerek oluşturulmuştur (T.C. Sağlık Bakanlığı, 2010). Formda kadınların AP bilgilerini sorgulayan toplam 20 soru (kadın kondomu cinsel yola bulaşan hastalıklardan korur, gebeliği önleyici hapların yan etkilerinden biri kilo artışıdır gibi) bulunmaktadır. Aile Planlaması Bilgi Formunun kapsam geçerliliğini sağlamak için uzman görüşü alınacak ve öneriler doğrultusunda gerekli düzenlemeler yapılacaktır. Formun içerik geçerliliği Polit ve Beck (2006)'in belirttiği gibi, Waltz ve Bausell (1981) tarafından geliştirilen İçerik Geçerliliği İndeksi (Content Validity Index =CVI)'ne dayalı olarak geliştirilecektir. Bu indekse göre uzmanlar her maddeyi "1" ile "4" arasında değişen puanlarla (1=Uygun değil, 2=Maddenin uygun şekle getirilmesi gerekir, 3=Uygun ancak küçük değişiklikler gerekir, 4=Çok uygun) değerlendirilecek ve her bir maddenin ölçme derecesini değerlendirmek üzere (3) ve (4) seçeneklerini işaretleyen uzmanların sayısı toplam uzman sayısına bölünerek her bir maddenin CVI değeri belirlenecektir. Her bir maddenin CVI değeri toplanıp formdaki madde sayısına bölünerek Aile Planlaması Bilgi Formunun CVI değeri hesaplanacak ve en az 0,80 olması durumunda formun içerik geçerliliğinin yeterli olarak değerlendirilecektir (Polit ve Beck, 2006).

Aile Planlaması Tutum Ölçeği: Örsal ve Kubilay tarafından 2007 yılında geliştirilmiş olup, üç alt boyutu bulunmaktadır. Ölçeğin "Toplumun Aile Planlamasına İlişkin Tutumları" alt boyutunda 15 soru, "Aile Planlama Yöntemlerine İlişkin Tutumlar" alt boyutunda 11 soru ve "Doğuma İlişkin Tutumlar" alt boyutunda 8 olmak üzere toplam 34 sorudan oluşmaktadır. Beşli likert tarzda olan bu ölçekte her madde 1'den 5'e kadar puanlanmakta ve toplamda en az 34, en fazla 170 puan

alınmaktadır. Ölçeğin cronbach alfa değeri 0,90 olup, madde ölçek korelasyon değerleri en düşük 0,31, en büyük 0,59 olarak bildirilmiştir. Ayrıca puan sayısı arttıkça güvenirlik katsayısı artmaktadır (Örsal ve Kubilay, 2007).

#### Verilerin Toplanması

İki grup için de kadınlarla tanışılarak araştırmanın amacı ve çalışma planı hakkında bilgi verilecektir. Çalışmaya katılmayı kabul eden kadınların sözlü ve yazılı onamları alınacaktır. İlk görüşmede Kişisel Bilgi Formu'nun birinci bölümü yüz yüze görüşme tekniğiyle doldurulacak olup, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği kadının kendi bildirimine göre doldurulacaktır. İlk görüşme sonlandırılmadan önce kadına üç ay sonra telefon ile aranılacağı, online anket formun gönderileceği ve bunun doldurulması gerektiği bilgisi verilecektir. İkinci görüşmede, Tanıtıcı Bilgi Formu'nun ikinci bölümü, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği online anket form doldurma yöntemi aracılığıyla doldurulacaktır.

#### Araştırmanın Uygulanması

#### Birinci aşama

- · Aile Sağlığı Merkez'ine bebeğinin bakım ve takibi için gelen, dahil edilme kriterlerine uyan, çalışmaya katılmaya gönüllü olan kadınlara çalışma hakkında bilgi verilecek ve çalışmaya katılmaya gönüllü olanlara "Bilgilendirilmiş Onam Formu" imzalatılacaktır.
- · Kişisel Bilgi Formu'nun birinci bölümü yüz yüze görüşme tekniğiyle doldurulacak olup, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği kadının kendi bildirimine göre doldurulacaktır. Bu süreçte araştırmacı tarafından kadınların mahremiyetine dikkat edilecektir.
- -Ardından her birinin üzerinde aile planlaması ile ilgili yazılı ve görsel mesajların bulunduğu iki paket hijyenik ped (bir paketin içinde 14 adet hijyenik ped olmak üzere toplam 28 adet) kadınlara teslim edilecektir. Birinci paketi ilk menstrual siklusunda, diğerini ise ikinci mestrual siklusunda kullanması söylenecektir.
- · Kadınların iletişim bilgileri alınacak, araştırmacı tarafından üç ay sonra iletişim kurulacağı, online anket formun gönderileceği ve bunun doldurulması gerektiği bilgisi verilecektir.

# İkinci aşama

- -Araştırmacı hijyenik pedler verildikten üç ay sonra kadın telefon ile iletişim kuracak ve kadının gönderilen online anket formu doldurması (Tanıtıcı Bilgi Formu'nun ikinci bölümü, Aile Planlaması Bilgi Formu ve Aile Planlaması Tutum Ölçeği) istenilecek.
- -Araştırmaya katılım sağlandığı için teşekkür edilecek ve veda edilecektir.

#### Araştırmanın Uygulama Akış Şeması

Aile Sağlığı Merkezi'ne bebeğinin bakım ve takibi için gelen kadınların araştırmaya dahil edilme kriterlerine uyup uymadığının değerlendirilmesi

Seçim kriterlerine uygun olan kadınların randomize olarak gruplara ayrılması

Kadınlara çalışma hakkında bilgi verilmesi ve kabul edenlerde yazılı ve sözlü onam alınması

#### Müdahale grubu

- Bilgilendirilmiş Onam Formu'nun imzalatılması,
- Veri toplama formunun birinci bölümü, Aile Planlaması Bilgi Formu ve Aile planlaması Tutum Ölçeği'nin doldurulması,
- İletişim bilgilerinin alınması,
- Üzerinde aile planlaması yöntemleri ile ilgili mesajlar yazan 2 paket (her pakette 14 adet olmak üzere toplam 28 adet) hijyenik ped verilmesi,
- İlk menstrual kanama bitiminden üç ay sonra iletişim kurulacağı bildirilmesi,
- Hijyenik pedler verildikten üç ay sonra veri toplama formunun ikinci bölümünün, Aile Planlaması Bilgi Formu ve Aile planlaması Tutum Ölçeği'nin doldurulması,
- Araştırmaya katılım için teşekkür sunulması ve veda edilmesi,

### Kontrol grubu

- Bilgilendirilmiş Onam Formu'nun imzalatılması,
- Veri toplama formunun birinci bölümünün,
   Aile Planlaması Bilgi Formu ve Aile
   planlaması Tutum Ölçeği'nin doldurulması,
- İletişim bilgilerinin alınması,
- İlk menstrual kanama bitiminden üç ay sonra iletişim kurulacağı bildirilmesi,
- Üç ay sonra veri toplama formunun ikinci bölümünün, Aile Planlaması Bilgi Formu ve Aile planlaması Tutum Ölçeği'nin doldurulması,
- Talep edenlere üzerinde aile planlaması yöntemleri ile ilgili mesajlar yazan 2 paket (her pakette 14 adet olmak üzere toplam 28 adet) hijyenik ped hediye edilmesi,
- Araştırmaya katılım için teşekkür sunulması ve veda edilmesi,

#### Randomizasyon

Çalışma, müdahale grubu ve kontrol grubu olmak üzere iki gruptan oluşacaktır. Çalışmada, dahil edilme kriterlerine uyan kadınların hangi grupta yer alacakları rastgele sayı üretme programı "Random Team Generator" adlı web sitesinden belirlenerek iki gruba ayrılacaktır. Böylece her kadının numarası ve grup numarası belirlenerek kaydedilecektir.

#### Körleme

Araştırmada müdahale grubunda yer alan kadınlara üzerinde yazılı ve görsel hijyenik ped vereceği için araştırmacıyı gruplara kör etmek mümkün değildir. Ancak katılımcıların hangi grupta yer alacağı "Random Team Generator" adlı web sitesinden belirleneceği için araştırmacının gruplara atama işlemi kör tutulacaktır. Kişisel Bilgi Formu'nun ikinci bölümü, Aile Planlaması Bilgi Formu ve

Aile Planlaması Tutum Ölçeği kadınların kendi bildirim yolu ile toplanacak ve araştırmacıların ölçek sonuçlarına kör olması sağlanacaktır. Verilerin analizi randomizasyon ve verilerin toplanması aşamalarında yer almayan üçüncü araştırmacı tarafından yapılmak körleme sağlanacaktır.

#### Değişkenler

Bağımlı değişkenler: Araştırmanın bağımlı değişkenlerini, Aile Planlaması bilgileri, Aile Planlaması Tutum puanı oluşturacaktır.

Bağımsız değişkenler: Araştırmanın bağımsız değişkenlerini, sosyo-demografik ve obstetrik özellikler oluşturacaktır.

#### Verilerin Analizi

Çalışmanın verileri Statistical Package for the Social Sciences 24 programı kullanılarak değerlendirilecektir. Tanımlayıcı istatistikler için, genelinde yüzde, normal dağılıma uygun olanlar için, aritmetik ortalama±standart sapma, uygun olmayanlar için ortanca ve minumum-maksimun değerler kullanılacaktır. Tüm veriler ilk önce, normal dağılıma uygunluk için Kolmogorov-Smirnov ile değerlendirilip, sonrasında normal dağılıma uygunluk durumuna göre analize alınacaktır. Verilerin analizinde, normal dağılıma uygun olanlar için student t testi, ANOVA testi, eşli iki örnek t testi, uygun olmayanlar için Mann-Whitney U, Kruskal Wallis testi, Wilcoxon testi, Friedman testi kullanılacaktır. Tip 1 hata düzeyi ise 0,05 olarak alınacaktır.

# Gönüllülerin (Olguların) Çalışmaya Katılmasına İlişkin Düzenlemeler

Gönüllülere araştırmanın amacı açıklanacak ve katılmayı kabul eden kadınların yazılı ve sözlü onamları alınacaktır. Veri toplama formlarını eksik dolduranlar ve araştırmanın herhangi bir aşamasında araştırmadan ayrılmak isteyenler araştırma dışı bırakılacaktır.

# Çalışmanın İzlenmesi ve Denetlenmesi

Çalışmanın veri toplama aşamasında ikinci araştırmacı tarafından veriler toplanacak ve birinci araştırmacı tarafından saha denetimi yapılacaktır. Araştırmacı, ebeler ile iletişim kurarak bebeğinin bakım ve takibi için ASM'ne gelecek kadınların randevu günlerini öğrenip o gün ASM'ne giderek araştırma verilerini toplanacaktır.

# Kullanılacak Malzemeler ve Saklama Koşulları ve Sorumluluklar

Aile Planlaması İle İlgili Mesajlar Yazan Hijyenik Ped: Hijyenik pedlerin üzerinde yazan bilgiler araştırmacılar tarafından hazırlanmış olup, aile planlaması yöntemlerinden hangilerine yer verileceği konusunda Türkiye Nüfus ve Sağlık Araştırması (TNSA) (2018)'ndan faydalanılmıştır. Türkiye Nüfus ve Sağlık Araştırması (2018) verilerine göre, 15-49 yaş aralığındaki halen evli kadınların %49'unun modern aile planlaması yöntemi, %21'inin geleneksel aile planlaması yöntemi kullandığı, kullanılan aile planlaması yöntemlerin ise sırasıyla; geri çekme (%20), kondom (%19), RİA (%14), tüpligasyon (%10), hap (%5) ve enjeksiyon (%1) olduğu bildirilmiştir (Hacettepe Üniversitesi Nüfus Enstitüsü, 2018). Bu veriler incelendiğinde, hijyenik ped üzerinde modern aile planlaması yöntemleri (hap, RİA, enjeksiyon, implant, kondom, diyafram, spermisit, tüpligasyon ve vazektomi) ile geleneksel aile planlaması yöntemlerinden geri çekme ve takvim yönteminin olması

gerektiğine karar verilmiştir. Aile planlaması yöntemlerine karar verildikten sonra eğitimin içeriğinin T.C. Sağlık Bakanlığı Ana Çocuk Sağlığı ve Aile Planlaması Genel Müdürlüğü tarafından 2010 yayınlanan rehber referans alınmıştır (T.C. Sağlık Bakanlığı, 2010). Bu rehberde, modern ve geleneksel aile planlaması yöntemleri ile ilgili basit, anlaşılır ve yalın bilgiler bulunmaktadır. Çalışmamızda, müdahale grubunda yer alan katılımcılara aile planlaması yöntemleri ile ilgili mesajlar yazan 15 adet hijyenik ped hazırlanmıştır. Mesajlar Microsoft word dosyasında hazırlanmış olup, yapışkan kağıt üzerine renkli çıktı alınacaktır. Alınan çıktılar pedlerin dış kılıfına yapıştırılacağı için sterilliği etkilenmeyecektir. Tüm kayıtlar 5 yıl süreyle sorumlu araştırmacı tarafından saklanacaktır.